CLINICAL TRIAL: NCT05619640
Title: The Potential Role of Receptor for Advanced Glycation End-Products, Serum, Krebs Von Den Lungen-6, and Surfactant Protein D as Prognostic Factors in Children With Severe Acute Respiratory Syndrome (SARS-CoV-2)
Brief Title: The Potential Role of sRAGE, KL-6, and SP-D as Prognostic Factors in Children With COVID-19
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gulsen Akkoc, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: 21/360
Record Dates: First submitted 2022-11-09; First posted 2022-11-17 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: SARS CoV 2 Infection; Alveolar; Injury; Children; Pneumonia, Viral
Keywords: soluble receptor for Advanced Glycation end products; Krebs von den Lungen-6; Surfactant protein D; Children; SARS CoV 2 Infection; Pneumonia
MeSH Terms: conditions — COVID-19; Wounds and Injuries; Pneumonia, Viral; Medullary cystic kidney disease 1; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 3-5 cc serum was obtained from participants. serum samples were stored at -80° C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: The study group divided into 3 groups according to COVID-19 WHO Clinical progression scale: Uninfected; No viral RNA detected
- Group 2: The study group divided into 3 groups according to COVID-19 WHO Clinical progression scale: Ambulatory mild disease Viral RNA detected but asymptomatic course, Symptomatic but not given any medication and Symptomatic given medication
- Group 3: The study group divided into 3 groups according to COVID-19 WHO Clinical progression scale: Hospitalized moderate disease Hospitalized but no oxygen therapy and Hospitalized and given oxygen by mask or nasal cannula

SUMMARY:
COVID-19 causes a wide spectrum of clinical illness, from upper respiratory symptoms to severe respiratory failure and death. Several plasma biomarkers -such as IL-6, C-reactive protein (CRP), D-dimer, the neutrophil-to-lymphocyte ratio, and ferritin, among others- have been studied as markers of disease severity and prognosis. Besides, as alveolar damage biomarkers such as Surfactant protein D (SP-D), Krebs von den Lungen-6 (KL-6), and soluble Receptor for Advanced Glycation end products (sRAGE) can be used in lung diseases as well as COVID-19 pneumonia. The investigators hypothesized that serum SP-D, KL-6 and sRAGE levels increases in the setting of COVID-19 pneumonia. In this prospective study the investigators aimed to determine the clinical value of serum KL-6, SP-D and sRAGE levels as a prognostic marker in children with COVID-19 patients. In the literature review, it has been determined that there is no study conducted or published in pediatric patients for this purpose, and it is aimed that our study will be a pioneer study on this subject.

DETAILED DESCRIPTION:
It aimed to determine the clinical value of serum KL-6, SP-D and sRAGE levels as a prognostic marker in children with COVID-19 patients.. This study was planned as a case-control study with patients hospitalized in the Haseki Training and Research Hospital Pediatric Infection Ward. A total of 150 children, including at least 30 patients in each group were included in the study. The study group was divided into three groups according to COVID-19 WHO clinical progression Scale: uninfected (Group 1), mild (Group 2) and moderate (group 3). In order to investigate the relationship between disease severity and alveolar damage, serum KL-6, SP-D and sRAGE levels and high sensitive C-reactive protein were measured. These biomarkers levels were compared between three groups.

ELIGIBILITY:
Inclusion Criteria:

1. Between 1 month-18 years old
2. SARS-CoV-2 PCR positive
3. Not having a chronic disease (cystic fibrosis, etc.)
4. Volunteering to participate in the study
5. Healty Control

Exclusion Criteria:

1. Having a chronic disease
2. Patients who could not be diagnosed with SARS-CoV-2 infection by laboratory and/or radiological examinations
3. Not volunteering to participate in the stud

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children and adolescents diagnosed as diagnosed SARS-CoV-2 infection and whose parents sign the informed consent from to participate the study
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Relationship between SARS-CoV-2 severity and alveolar damage biomarker levels | baseline
  Serum samples were obtained from all patients on admission. The data set divided into three groups according to COVID-19 WHO Clinical progression scale. The Surfactant protein D, Krebs von den Lungen-6, high sensitive C-reactive protein and soluble receptor for Advanced Glycation end products levels were determined by using ELISA kits. These biomarker levels were compared between three groups by using Kruskal-Wallis test and Tukey post test for multiple comparisons.

CONTACTS AND LOCATIONS:
Overall Officials: Gulsen Akkoc, M.D., Study Director — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The IPD are available from the principal investigator upon reasonable request

REFERENCES:
- [Background] WHO Working Group on the Clinical Characterisation and Management of COVID-19 infection. A minimal common outcome measure set for COVID-19 clinical research. Lancet Infect Dis. 2020 Aug;20(8):e192-e197. doi: 10.1016/S1473-3099(20)30483-7. Epub 2020 Jun 12. PMID 32539990
- [Result] Determann RM, Royakkers AA, Haitsma JJ, Zhang H, Slutsky AS, Ranieri VM, Schultz MJ. Plasma levels of surfactant protein D and KL-6 for evaluation of lung injury in critically ill mechanically ventilated patients. BMC Pulm Med. 2010 Feb 16;10:6. doi: 10.1186/1471-2466-10-6. PMID 20158912
- [Result] Kommoss FKF, Schwab C, Tavernar L, Schreck J, Wagner WL, Merle U, Jonigk D, Schirmacher P, Longerich T. The Pathology of Severe COVID-19-Related Lung Damage. Dtsch Arztebl Int. 2020 Jul 20;117(29-30):500-506. doi: 10.3238/arztebl.2020.0500. PMID 32865490
- [Result] Sivapalan P, Bonnesen B, Jensen JU. Novel Perspectives Regarding the Pathology, Inflammation, and Biomarkers of Acute Respiratory Distress Syndrome. Int J Mol Sci. 2020 Dec 28;22(1):205. doi: 10.3390/ijms22010205. PMID 33379178